CLINICAL TRIAL: NCT04827199
Title: Safety and Clinical Performance Study of the ARTUS® Artificial Urinary Sphincter (AUS) for the Treatment of Stress Urinary Incontinence (SUI) Due to Intrinsic Sphincter Deficiency
Brief Title: Safety and Clinical Performance Study of the ARTUS® Artificial Urinary Sphincter (AUS)
Acronym: DRY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Myopowers Medical Technologies France SAS (Industry)
Collaborators: EVAMED (Other); Affluent Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRY; CIV-CZ-22-01-038768 (Other: EUDAMED)
Record Dates: First submitted 2021-03-09; First posted 2021-04-01 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Stress Urinary Incontinence
Keywords: Artificial Urinary Sphincter
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: The subjects will be implanted with the ARTUS® medical device and then be followed up for 10 years post-implant, with the primary endpoints measured at 3-month post-device activation visit.
  As there is no comparator, there is no randomization and no blinding in the study.
  Clinical performance outcomes will be measured for each subject at baseline (before implantation) and post-implantation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARTUS® (Experimental): The subjects will be implanted with the experimental medical device ARTUS® Artificial Urinary Sphincter (AUS) during the surgical procedure and will be trained to the use of the Remote Control to control themselves the micturition.
  Interventions: Device: Artificial Urinary Sphincter implantation

INTERVENTIONS:
Device: Artificial Urinary Sphincter implantation — Device preparation (recharge, settings, pairing) Patient preparation Calibration procedure (to verify the device is in full working prior to implantation)
  Implantation procedure which includes:
  * Perineal approach and bulbar urethral dissection
  * Inguinal approach
  * Cuff implantation around the urethra
  * Transmission cable passing
  * Surgery test procedure
  * Implantation of the Control Unit
  * Closure of the inguinal incision
  * Closure of the perineal incision
  * "Implant disabled mode" activation

SUMMARY:
This clinical investigation is designed as an interventional, prospective, non-randomized, open-label, single arm, multicentric and international study for obtaining CE marking.

The study will be the first performed with the ARTUS® medical device aiming to assess safety and performance and will be composed of three phases:

* pilot phase (with safety analysis on the 10 first included subjects in 3 investigational sites),
* pivotal phase (in up to 16 investigational sites with a follow-up until the 12-month post-device activation visit, including an interim analysis at 3-month post-device activation visit on performance and safety),
* long-term phase (with a long-term follow-up until 10 years post implantation in up to 16 investigational sites).

The objectives is to assess safety and clinical performance of the ARTUS® for the treatment of Stress Urinary Incontinence at short and long-term.

ELIGIBILITY:
Inclusion Criteria:

1. Male subject between 18 and 80 years (inclusive) of age at the time of consent signature
2. Subject with persistent urinary incontinence, defined as >12 months
3. Subject with severe Stress Urinary Incontinence, defined as a mean value of 3 consecutive 24-hour Pad Weight Test > 75 grams
4. Subject willing and able to provide written informed consent
5. Subject willing and able to comply with all clinical study requirements, including the ability to independently operate the device remote control
6. Subject willing and able to comply with follow-up visits
7. Subject having understood and accepted to be unable to proceed to an MRI examination after the surgical procedure due to the non-MRI compatibility of the device
8. Subject having signed the informed consent

Exclusion Criteria:

1. Subject with documented neurological bladder or history of neurological disease liable to interfere with urinary symptoms
2. Subject with history of Artificial Urinary Sphincter or male sling implantation
3. Subject with history of pelvic radiotherapy
4. Subject with history of Artificial Urinary Sphincter-related urethral erosion
5. Subject with history of urethral fistula
6. Subject with history of bladder tumour
7. Subject with severe urethral stenosis
8. Subject with urge incontinence due to hyperactive bladder not adequately controlled by drug therapy
9. Subject with severe congenital or acquired haemorrhagic disease, haemophilia, or another coagulopathy
10. Subject under anti-coagulation or anti-platelet medication that cannot be discontinued at least 5 days prior to surgery and restarted at least 5 days after surgery
11. Subject with currently active infection, including urinary tract infection
12. Subject with severe renal failure or obstructive pathologies of the upper urinary tract with severe renal failure
13. Subject with a current vesicourethral reflux
14. Subject with congenital or acquired immunodeficiency, including those who are immunocompromised or immunosuppressed
15. Subject with bladder or urethral foreign body or calculus
16. Subject with allergy to any components of the device
17. Subject deprived of liberty by administrative or judicial decision or under legal guardianship
18. Subject having a Body Mass Index (BMI) > 40
19. Subject with post void residual volume greater than 200 mL, within the past 6 months
20. Subject with uncontrolled diabetes, defined as HbA1c > 9.0%, within the past 6 months
21. Subject with history of recurrent bladder stones or history of failed bladder stone treatment within the past 12 months
22. Subject currently enrolled or plans to participate in another investigational study of a drug, biologic, or medical device from the point of enrolment through the 12 months post device activation period
23. Subject who underwent any surgical procedure in the last 3 months, or with planned surgical procedure within the next 3 months
24. Subject who is unwilling or deemed by the Investigator to be unwilling to comply with the Clinical Investigation Plan, or subject with a history of non-compliance
25. Subject unable to understand and sign the ICF in absence of legal representative
26. Subject with a lack of capacity to consent
27. Subject unable to read and write
28. Subject in emergency situation

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Change in the 24-hour Pad Weight Test | 3 months post-device activation
  Proportion of subjects with at least 50% reduction in 24-hour Pad Weight Test at 3 months post-device activation compared to baseline.

SECONDARY OUTCOMES:
Adverse events (including adverse device effect) occurred from the implantation to the 10-year follow-up period | Implantation, 6 weeks, 8 weeks and 3 months post-op, 3 months, 6 months, 12 months post-device activation, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years post-op
  All adverse events (including adverse device effect) occurred from the implantation to the 10-year follow-up period, with their occurrence, severity and nature.
  All adverse events will be analysed and classified using the Clavien-Dindo classification grading system
Revision rate | Implantation, 6 weeks, 8 weeks and 3 months post-op, 3 months, 6 months, 12 months post-device activation, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years post-op
  Proportion of subjects who have been concerned with a revision between the implantation and each visit (or scheduled visit date), until the 10-year follow-up period
Explantation rate | Implantation, 6 weeks, 8 weeks and 3 months post-op, 3 months, 6 months, 12 months post-device activation, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years post-op
  Proportion of subjects who have been concerned with an explantation of the medical device between the implantation and each visit (or scheduled visit date), until the 10-year follow-up period
Renal function | Baseline, Implantation, discharge, 3 months, 6 months, 12 months post-device activation, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years post-op
  Assessed using the serum creatinine
Pain assessed by numeric rating scale | Implantation, 6 weeks, 8 weeks and 3 months post-op, 3 months, 6 months, 12 months post-device activation, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years post-op
  Pain assessed using a 10-point numeric rating scale where 0 is no pain and 10 is the worst pain imaginable
Voided urine assessed with uroflowmetry | Baseline, 3, 6 and 12-month post-device activation, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years post-op
  Voided urine assessed with uroflowmetry per unit of time (mL/s)
Voided volume assessed with uroflowmetry | Baseline, 3, 6 and 12-month post-device activation, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years post-op
  Voided volume assessed with uroflowmetry in mL and maximum flow rate (Qmax)
Maximum flow rate assessed with uroflowmetry | Baseline, 3, 6 and 12-month post-device activation, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years post-op
  Maximum flow rate assessed with uroflowmetry (Qmax)
Bladder drainage | Baseline, 3, 6 and 12-month post-device activation, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years post-op
  Assessed using post-void residual volume
Usability assessed by a 5-point scale | Implantation
  Usability assessed by a 5-point scale from 1 (strongly agree) to 5 (strongly disagree)
Device deficiencies occurred from the implantation to the 10-year follow-up period | Implantation, 6 weeks, 8 weeks and 3 months post-op, 3 months, 6 months, 12 months post-device activation, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years post-op
  Device deficiencies occurred from the implantation to the 10-year follow-up period with their occurrence and nature.
Change in the 24-hour Pad Weight Test | Baseline, 3, 6 and 12-month post-device activation
  24-hour Pad Weight Test
Reduction in the 24-hour Pad Weight Test | Baseline, 6 and 12-month post-device activation
  Proportion of subjects with at least 50% reduction in 24-hour Pad Weight Test
Pad Usage | Baseline, 3, 6, and 12-month post-device activation visit,2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years post-op
  Number of pads/day
Urinary symptoms assessed with ICIQ-MLUTS subscales | Baseline, 3, 6, and 12-month post-device activation visit, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years post-op
  Urinary symptoms assessed with ICIQ-MLUTS subscales :
  * Voiding symptoms subscales from 0 (no symptom) to 20
  * Incontincence symptoms subscales from 0 (no symptom) to 24
Urinary incontinence Quality of Life assessed with ICIQ-LUTSQoL questionnaire | Baseline, 3, 6, and 12-month post-device activation visit, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years post-op
  Urinary incontinence Quality of Life assessed with ICIQ-LUTSQoL questionnaire score from 19 to 76 with greater values indicating increased impact on quality of life
General Quality of Life assessed with EQ-5D-5L questionnaire | Baseline, 3, 6, and 12-month post-device activation visit, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years post-op
  The EQ-5D-5L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) of 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Sexual Quality of Life assessed with the Male Sexual Health Questionnaire (MHSQ) | Baseline, 3, 6, and 12-month post-device activation visit, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years post-op
  The MSHQ is a 25-item self-administered questionnaire. It encompasses 3 scales: Erection scale (3 items), Ejaculation scale (7 items), Satisfaction scale (6 items), and 9 additional items addressing sexual activity, time since last sexual encounter, level and changes in sexual activity, and bother associated with sexual dysfunction. Response options consist of dichotomous (Yes/No) scales, as well as 5 and 6- point likert scales.
  Scores by dimension:
  * Erection scale: 0-15 (higher score =higher sexual functioning)
  * Ejaculation scale: 1-35 (higher score =higher sexual functioning)
  * Satisfaction scale: 6-30 (higher score =higher level of satisfaction)
Subject usability assessed by a 5-point scale | 3, 6, and 12-month post-device activation visit, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years post-op
  Subject usability questionnaire completed by the subject from 1 (strongly agree) to 5 (strongly disagree)
Subject satisfaction assessed by the PGI-I | 3, 6, and 12-month post-device activation visit, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years post-op
  Subject satisfaction assessed by the PGI-I questionnaire which includes a unique 7-point scale to describe how the post-operative condition is now, compared with how it was before the surgery and where 1 = Very much better and 7 = very much worse
Subject satisfaction assessed by 5-point scale | 3, 6, and 12-month post-device activation visit, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years post-op
  Subject satisfaction assessed by the question "Are you satisfied with the use of ARTUS" with the 5-point scale answers where 1 = strongly agree and 5 = Strongly disagree
Subject recommendation assessed by 5-point scale | 3, 6, and 12-month post-device activation visit, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years post-op
  Subject recommendation assessed by the question "Would you recommend ARTUS to a friend" with the 5-point scale answers where 1 = strongly agree and 5 = Strongly disagree
Investigator usability assessed by a 5-point scale | Device activation visit (6 weeks post-operative visit), 3 months post-device activation
  Investigator usability questionnaire completed by the investigator from 1 (strongly agree) to 5 (strongly disagree)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Zachoval, Pr, Principal Investigator — Thomayerova nemocnice; Marion Melot, Study Director — Myopowers Medical Technologies France SAS
Locations (3):
- Thomayer hospital, Prague, Czechia
- Spain (2):
  - Hospital Germans Trias i Pujol, Barcelona, Badalona
  - Hospital Clinico San Carlos, Madrid

IPD SHARING:
Plan to Share IPD: No